CLINICAL TRIAL: NCT02790489
Title: Valedia Dietary Supplement Tolerance Study Based on Blood, Urinary and Hemodynamic Biological Parameters
Brief Title: Tolerance Study of the Dietary Supplement Valedia
Acronym: ECPH1-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Centre d'Investigation Clinique INSERM 501, Clermont-Ferrand, France (Unknown); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A01864-45
Record Dates: First submitted 2016-05-17; First posted 2016-06-06 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valedia (Experimental): Dose 1 : 2,5 g (4 capsules) Valedia per day during 4 weeks Dose 2 : 5 g (8 capsules) Valedia per day during 4 weeks 2 weeks (wash-out period) between the 2 doses
  Interventions: Dietary Supplement: Valedia

INTERVENTIONS:
Dietary Supplement: Valedia

SUMMARY:
The objectives of this clinical study are to determine the tolerance of dietary supplement Valedia (blend of plant extracts) through the evaluation of several parameters :

* Various blood biological parameters for tolerance (preprandial): blood glucose, insulin, fructosamine, total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol, oxidized LDL, us-CRP, creatinine, ASAT, ALAT, gGT, phosphatase alcaline, bilirubine, urea.
* Urinary parameters: urea, creatinine.
* Hemodynamic parameters: heart rate and blood pressure.
* Cardiac function: ECG.
* Weight.

ELIGIBILITY:
Main Inclusion Criteria:

* 25 <= BMI < 30 kg.m2

Main Exclusion Criteria:

* ASAT <= 1,55 microkat/L
* ALAT <= 1,70 microkat/L
* gGT <= 2,55 microkat/L
* 55 <= Creatinine <= 104 micromol/L (+- 10%)
* Bilirubin < 17,1 micromol/L (+- 10%)
* 1,7 <= Urea <= 8,3 mmol/L (+- 10%)
* us-CRP <= 5 mg/L (+- 10%)
* 0,70 <= Fasting glycemia <= 1,25 g/L (+- 10%)
* HbA1c <= 6%
* Medications for diabetes and/or dyslipidemia

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Effect on urine urea | 10 weeks
  Urine urea
Effect on urine creatinine | 10 weeks
  Urine creatinine
Effect on fasting glycemia | 10 weeks
  Fasting blood glucose
Effect on insulin | 10 weeks
  Plasma insulin
Effect on fructosamine | 10 weeks
  Blood fructosamine
Effect on total cholesterol | 10 weeks
  Blood total cholesterol
Effect on HDL cholesterol | 10 weeks
  Blood HDL cholesterol
Effect on LDL cholesterol | 10 weeks
  Blood LDL cholesterol
Effect on triglycerides | 10 weeks
  Blood triglycerides
Effect on oxidized LDL cholesterol | 10 weeks
  Blood oxidized LDL cholesterol
Effect on inflammation | 10 weeks
  Blood us-CRP
Effect on AST | 10 weeks
  Blood AST
Effect on ALT | 10 weeks
  Blood ALT
Effect on gamma GT | 10 weeks
  Blood gamma GT
Effect on alkaline phosphatase | 10 weeks
  Blood phosphatase alkaline
Effect on bilirubin | 10 weeks
  Blood bilirubin
Effect on cardiac function | 10 weeks
  ECG

SECONDARY OUTCOMES:
The response during an oral glucide tolerance test after a standardized breakfast | 10 weeks
  Oral glucose tolerance test (after a standardized breakfast) with glycemia and insulinemia measurements (-10 min, -5 min, +15 min, +30 min, +45 min, +60 min, +90 min, +120 min, arrival at center in fasting state)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien L Peltier, PhD, Study Director — Valbiotis
Locations (1):
- Centre d'Investigation Clinique, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes